CLINICAL TRIAL: NCT00558649
Title: A Pilot, Controlled, Comparative and Single Blinded Study to Evaluate the Safety and Immunogenicity of Low Dose Flu Vaccines Administered Intradermally Using Microneedle Injectors as Compared With Standard Dose Intramuscular Flu Vaccines as Reference.
Brief Title: A Pilot Study to Evaluate the Safety and Immunogenicity of Low Dose Flu Vaccines
Acronym: NANOVAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NanoPass Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NP39; EudraCT number 2007-001160-77
Record Dates: First submitted 2007-05-27; First posted 2007-11-15 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2007-11

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; fluarix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Low dose flu vaccine delivered intradermally using microneedles
  Interventions: Biological: Flu Vaccine (FLUARIX®)
- 2 (Experimental): Medium dose flu vaccine delivered intradermally using microneedles
  Interventions: Biological: Flu Vaccine (FLUARIX®)
- 3 (Active Comparator): Standard dose flu vaccine delivered intramuscularly with a regular needle
  Interventions: Biological: Flu Vaccine (FLUARIX®)

INTERVENTIONS:
Biological: Flu Vaccine (FLUARIX®) — Influenza Virus Vaccine, FLUARIX®, 2006-2007 Formula

SUMMARY:
The purpose of this study is to determine whether low dose flu vaccines delivered with microneedles into the skin (intradermally) are effective.

DETAILED DESCRIPTION:
Influenza vaccination is the primary method for preventing influenza and its severe complications. Previous clinical studies demonstrated that delivery of vaccines intradermally (into the skin) can achieve good efficacy even with lower doses of the vaccine.

Comparison: Low dose flu vaccine delivered intradermally with a microneedle device compared to the standard dose flu vaccine delivered intramuscularly (into the muscle) with a regular needle.

ELIGIBILITY:
Inclusion Criteria:

* Signed an Informed Consent
* No previous immune-related disease

Important Exclusion Criteria:

* Significant illness within the previous 4 weeks
* Subjects who have received an influenza vaccine within the previous 6 months
* An active viral diseases
* Pregnant or nursing women
* Any known contraindication to the study vaccine or vaccine ingredients

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2007-05; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Van Damme, MD, PhD, Principal Investigator — Center for the Evaluation of Vaccination, University of Antwerp